CLINICAL TRIAL: NCT01546844
Title: Use of Mobile Health Technology as an Intervention for Type II Diabetes Self-Management
Brief Title: Mobile Health Technology as an Intervention for Diabetes Self-Management
Acronym: Care4Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: HealthInsight (Other)
Collaborators: Center for Technology and Aging (Unknown); Voxiva (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Care4Life Grant
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Type II Diabetes Mellitus
Keywords: SMS; text; text messages; text messaging; diabetes; diabetes mellitus; type II diabetes; type II diabetes mellitus; type 2 diabetes; type 2 diabetes mellitus; Beacon
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care4Life (Experimental): Text message and online interactive component to help patients with self-management.
  Interventions: Other: Participation in Care4Life
- Standard of Care (No Intervention): Patients enrolled in this arm will receive their normal standard of care from their physician for treatment of type II Diabetes Mellitus.

INTERVENTIONS:
Other: Participation in Care4Life — Text message service to aid patients with self-management of type II Diabetes Mellitus. Includes online access to patient data and management of health goals.
  Other Names: Voxiva
  Arms: Care4Life

SUMMARY:
This purpose of this is study is to evaluate the effectiveness of an interactive mobile health information service, Care4Life, in supporting patient self-management of Type II Diabetes Mellitus.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of an interactive mobile health information service, Care4Life, in supporting patient self-management through its ability to facilitate patient education, behavior change, and improved adherence with standard care practices. The study population comprises adults who have been diagnosed with Type 2 diabetes mellitus (DM) and a hemoglobin A1c (HbA1c) test above 8% in the past year. All members of the study population are treated at primary care clinics under the auspices of the Utah Beacon Community Program, which aims to improve health through use of health information technology. We will compare outcomes in two groups within this population: patients with DM who enroll in Care4Life (in addition to receiving standard care) to patients with DM who receive standard care from their physician. We will compare these groups both within the clinic and at an aggregated, overall level.

This study relies on the use of information and communications technology (ICT) in supporting patient-empowerment strategies. Features of successful diabetes care programs for improving adherence to standards of care, such as the use of diabetes self-management education, checklists that mirror guidelines, and automated reminders are well suited to delivery using an interactive mobile health platform.

Research Questions

This study will evaluate the efficacy of the Care4Life mHealth program by:

1. Evaluating if a short message service via cell phone texting (SMS) protocol will lead to improvements in clinical, utilization and satisfaction outcomes for patients with DM compared to patient who receive standard care.
2. Evaluating if an SMS protocol can be readily adopted by an adult population in both urban and rural areas with a time-consuming chronic illness.

Targeted outcomes include:

1. Improved measures of diabetes control, demonstrated as HbA1c percentage levels ≤ 8%; improved blood pressure (BP) control, demonstrated as BP ≤ 140/90 millimeters mercury (mm Hg); and lower body mass index (BMI) among users of the SMS-based tool.
2. Improved knowledge of self-care and disease management practices among adult patients with diabetes treated in Beacon clinics in the Salt Lake Metropolitan Statistical Area (Salt Lake, Tooele, and Summit counties).
3. Dissemination of results and proof of concept with the broader healthcare community in Utah.

The mobile centric diabetes support service at the center of our study is Voxiva's Care4Life platform, which is an interactive mobile application designed to educate participants, encourage behavior change and promote adherence to their prescribed DM treatment protocol. It includes a series of SMS-based tools that have been developed in collaboration with the Instituto Carso de la Salud, located in Mexico. The service sends content relevant to the target participants and their standard treatment protocol. Care4Life delivers an individually tailored diabetes education and management plan based on data that are collected from patients at enrollment and added to the participant's personal health profile.

The SMS protocol draws on the experience of a number of interventions that have been independently studied and shown to improve health outcomes. Care4Life functionality consists of the following components: (1) a diabetes diary that can be used to develop a history of glucose levels and trigger alerts and feedback based on the participant's results; (2) health education with content tailored to the participant's health profile; (3) medication adherence reminders and monitoring; (4) medical appointment reminders; (5) a database that allows a participant to record and monitor her/his weight, BMI, blood pressure and laboratory results; and (6) a health portal that allows a participant to review his/her data, obtain advice and guidance based on the information entered, and manage his/her preferences.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory test for HbA1c ≥ 8% within the past year
* Clinical diagnosis of DM
* Age > 18 years old
* Patient in a Beacon clinic
* Cell phone ownership or willingness to acquire a cell phone capable of receiving and sending SMS messages
* Women who are not pregnant

Exclusion Criteria:

* Failure to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c - In control, over time. | 3, 6, 9, and 12 months
  Hemoglobin A1c - In control as assessed by laboratory results of blood draw taken from patient's clinic. In control means a result of <9%.

SECONDARY OUTCOMES:
Change in Blood Pressure Control over time | 3, 6, 9, 12 months
  Improved blood pressure (BP) control as demonstrated as BP ≤ 140/90 millimeters mercury (mm Hg)
Change in BMI over time | 3, 6, 9, 12 months
  Lower body mass index (BMI) among users of the SMS-based tool.
Disease Management | 12 months
  Improved knowledge of self-care and disease management practices among adult patients with diabetes treated in Beacon clinics in the Salt Lake Metropolitan Statistical Area (Salt Lake, Tooele, and Summit counties).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Woolsey, MD, Principal Investigator — HealthInsight; Korey Cappoza, MPH, Study Director — HealthInsight
Locations (30):
- United States (30):
  - Coalville Health Center, Coalville, Utah
  - Pioneer Comprehensive Medical, Draper, Utah
  - Holladay Family Practice, Holladay, Utah
  - Olympus Clinic, Holladay, Utah
  - Exodus Healthcare - Main Office - Magna, Magna, Utah
  - Community Health Centers Inc. - 72nd Street Clinic, Midvale, Utah
  - Park City Healthcare, Inc., Park City, Utah
  - Riverton Family Health Center, Riverton, Utah
  - Granger Medical-Riverton, Riverton, Utah
  - Wasatch Homeless Health Care - 4th Street Clinic, Salt Lake City, Utah
  - Alpine Internal Medicine, Salt Lake City, Utah
  - HealthInsight, Salt Lake City, Utah
  - Central City Community Health Center Health First Family Medicine, Salt Lake City, Utah
  - Evolutionary Healthcare, Llc, Salt Lake City, Utah
  - Health Clinic Of Utah - SLC, Salt Lake City, Utah
  - Stephen D. Ratcliffe Community Health Center, Salt Lake City, Utah
  - Jordan Ridge Family Medicine, Salt Lake City, Utah
  - Utah Healthcare Institute - St. Mark's Family Medicine, Salt Lake City, Utah
  - Utah Physicians Care Centers - St Mark's Internal Medicine, Salt Lake City, Utah
  - Wasatch Internal Medicine, Salt Lake City, Utah
  - Barbara E. Rizzardi, M.D., Sandy City, Utah
  - Copperview Medical Center, Llc, South Jordan, Utah
  - Community Health Centers Inc. - Oquirrh View, Taylorsville, Utah
  - Advanced Practice Medical Clinic, Tooele, Utah
  - Valley Family Medicine, Tooele, Utah
  - Granger Medical - Jordan Medical Arts, West Jordan, Utah
  - Jordan Meadows Medical Center, West Jordan, Utah
  - Granger Medical Clinic Inc. - Main Office, West Valley City, Utah
  - Kathryn Allen, MD, West Valley City, Utah
  - West Valley Family And Preventive Medicine, West Valley City, Utah